CLINICAL TRIAL: NCT03248661
Title: Assessing Repeat Annual FIT Screening for Colo-Rectal Cancer (CRC)
Brief Title: Assessing Repeat Fit Testing for CRC
Acronym: ARFT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Richard Crosby (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Richard Crosby, PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 14-0662-P3H
Record Dates: First submitted 2015-07-24; First posted 2017-08-14 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-01

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention media condition (Experimental): monthly social media contact will be used to keep people connected to the idea of completing a second screening test 12 months after their last one.
  Interventions: Behavioral: Now I'm Telling You
- control condition (No Intervention): this group will receive only a standard reminder for the annual repeat test, one month before the test due date

INTERVENTIONS:
Behavioral: Now I'm Telling You — Messages will be sent trough Facebook, Twitter, Instagram, e-mail, texting or other electronic/social media specified by study volunteers.
  Arms: Intervention media condition

SUMMARY:
This study will randomly assign 220 men and women to either a social media intervention or a standard reminder system to have a repeat screening test for colo-rectal cancer.

DETAILED DESCRIPTION:
Only persons initially screening by FIT (through a Rural Cancer Prevention Center service program) will be eligible for study participation. The objective is to test a social media-based intervention designed to promote annual repeat colo-rectal cancer screening using the Fecal Immunochemical Test (FIT) among person who have taken the FIT test once before. 220 men and women (50 to 75 years of age) will be recruited and randomly assigned to either the intervention condition (monthly social media contact) or a control condition (standard of care reminder for repeat testing one month before the annual test is due). The dependent variable will be whether volunteers requested and retuned a FIT kit with 60 days of the annual due date (one year from their initial screening).

ELIGIBILITY:
Inclusion Criteria:

* must have completed and returned an initial FIT kit to us as part of a Rural Cancer Prevention Center service program to the community

Exclusion Criteria:

* visible blood in stool or prior diagnosis of cool-rectal cancer

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is a received completed FIT kit within 15 months after the participant received results from the original FIT test | 15 months
  the endpoint is a received completed FIT kit

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States